CLINICAL TRIAL: NCT01990495
Title: Exercise to Prevent Muscle Mass and Functional Loss in Elderly Dialysis Patients
Acronym: PERFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E0915-R
Record Dates: First submitted 2013-10-30; First posted 2013-11-21 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Disease
Keywords: Renal failure; Exercise testing; Exercise training; Protein signaling; Skeletal muscle
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise vs. usual care (Active Comparator): The study involves two arms randomized to exercise and usual care groups
  Interventions: Other: Exercise training; Other: Usual Care
- Usual care (Active Comparator): This group will be randomized to receive usual clinical care. No other interventions will be assigned to this group.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Exercise training — Subjects will participate in a center-based and home exercise training program for 3 months.
  Arms: Exercise vs. usual care
Other: Usual Care — This group will serve as control subjects. They will receive only usual clinical care.

SUMMARY:
The majority of individuals with advanced ESRD have reduced exercise capacity in part due to decreased muscle mass. This leads to a reduced ability to perform daily activities, a greater incidence of falls, and a reduced quality of life. The mechanisms responsible for the loss of muscle mass in ESRD are not understood very well. This study is designed to determine the effectiveness of an exercise program on improving muscle mass, exercise capacity and quality of life in persons with ESRD. In addition, the study will attempt to better understand why muscle loss occurs in people with ESRD, the influence exercise has on these mechanisms, and whether the response to exercise can be enhanced with nutrient supplementation.

DETAILED DESCRIPTION:
Elderly patients comprising half the end-stage renal disease (ESRD) population, are especially vulnerable to loss of muscle mass, strength and function, changes that lead to frailty and increased morbidity and mortality. Many factors contribute to the decline in muscle mass and function in the elderly uremic and apart from aging and co-morbid conditions, wasting is worsened by inactivity. Studies in maintenance hemodialysis (MHD) patients have shown that exercise (EX), including endurance, resistance or combined, can counteract the loss of muscle mass and function. However most studies have not specifically targeted the elderly, involved small numbers or lacked controls and the impact on long-term outcome is unknown. Nevertheless, despite substantial evidence indicating that EX is beneficial and low cost, EX is not part of the routine care of MHD patients. In contrast EX is regarded as standard of care for the wasted elderly and also cardiac patients. Some protection against uremic muscle wasting can also be afforded by an adequate protein-calorie intake. Amino acids (AA) from this source serve as substrates for protein synthesis (PS) and also directly activate the mTOR signaling pathway stimulating PS. In normal subjects if AA are ingested at the time of resistance EX, anabolic signaling and PS is enhanced and this leads to increases in muscle mass. Whether the EX and AA stimulated signaling response is intact in elderly MHD patients is unknown and there is little information about the cellular processes invoked. Taking this all together, the investigators plan to test the hypothesis that a home-based EX program, effective in cardiac patients, will improve cardiopulmonary function and muscle mass and function in elderly MHD patients. Also, in a pilot study the investigators will examine whether a protein supplement acutely enhances EX stimulated anabolic signaling. Functionally impaired MHD subjects aged 65-80 yrs are randomized into 2 groups of 30 each, one undergoing EX and the other usual care. After 3 months, half in each group receive a one-time protein-calorie supplement or placebo during an acute bout of EX and muscle biopsied for examining the signaling response. Assays at baseline and at 3 months include cardiopulmonary function, muscle strength and function, body composition by DEXA, thigh muscle volume and composition by CT, quality of life (QOL) and cognitive function, and nutritional, inflammatory, lipid and biochemical status and morphologic and molecular analysis of biopsied muscle. The investigators anticipate that home-based EX will counteract muscle wasting, enhance cardiopulmonary and muscle function and QOL, and reduce surrogate markers of long-term outcome. New insights into the mechanisms whereby EX and nutrients induce an anabolic response in muscle of elderly uremics will be provided and may serve as a basis for devising strategies to counteract loss of muscle mass and function. Finally, the investigators anticipate that the EX program will be "user friendly" and may thus form a part of the routine care of elderly and perhaps younger MHD patients. If short-term benefits are evident from this study in elderly MHD patients, it could form the basis for a comprehensive long-term outcomes study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 55-80 years undergoing maintenance hemodialysis (MHD) for at least three months and without other active/uncontrolled disease will be studied.
* Exercise and usual care groups will be matched by age, body mass index (BMI), MHD duration, and protein intake using a stratified randomization approach.
* Subjects will be required to be in the peak VO2 range of 10 to 20 ml/kg/min, equivalent to moderate functional impairment in patients with heart failure.
* Subjects will be required to have dialysis treatment for >3 months with an average Kt/V 1.2, and be able to perform exercise safely.

Exclusion Criteria:

* Current activity > 2 hrs/wk of moderate intensity exercise, temporary vascular access, uncontrolled diabetes mellitus, active vasculitis, active autoimmune disease, malignancy, severe obesity (BMI > 35), alcoholism or other recreational drug use, unstable cardiac disease (abnormal exercise test, angina, uncontrolled arrhythmias or myocardial infarction within three months), peripheral vascular disease (claudication with exercise), lung, liver or intestinal disease, those who are medically unstable and subjects who have received anabolic, catabolic or cytotoxic medications in the past 3 months.
* The investigators will also exclude subjects with excessive previous exposure to radiation.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Neil Myers, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Myers J, Chan KN, Chen Y, Lit Y, Massaband P, Kiratli BJ, Tan JC, Rabkin R. Association of physical function and performance with peak VO2 in elderly patients with end stage kidney disease. Aging Clin Exp Res. 2021 Oct;33(10):2797-2806. doi: 10.1007/s40520-021-01801-6. Epub 2021 Mar 8. PMID 33686542

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: The study involves two arms randomized to exercise and usual care groups
  Exercise training: Subjects will participate in a center-based and home exercise training program for 3 months.
  Usual Care: This group will serve as control subjects. They will receive only usual clinical care.
Period: Overall Study
Arm/Group | Exercise | Usual Care
Started | 18 | 19
Completed | 13 | 15
Not Completed | 5 | 4
Not completed — Physician Decision | 5 | 4

BASELINE CHARACTERISTICS:
Population: Chronic kidney disease on maintenance hemodialysis.
Groups:
- Exercise: Subjects will participate in a center-based and home exercise training program for 3 months.
- Total: Total of all reporting groups
Arm/Group | Exercise | Usual Care | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 10 | 13 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.6) | 66.2 (6.7) | 66.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximal Oxygen Uptake
Description: The overall primary outcome for the study is maximal oxygen uptake. Maximal oxygen uptake is the amount of oxygen consumed by the body during maximal exercise. It is the gold standard expression for exercise capacity.
Time Frame: 3 months
Population: Chronic kidney disease
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 15
ml/kg/min | 14.5 (3.3) | 15.1 (3.3)

2. Secondary Outcome: Biopsy of the Quadriceps Muscle.
Description: The biopsy procedures will permit the measurement of the percentage of type 1 fibers in the quadriceps muscle.
  The biopsy procedures will also be used to quantify protein signaling, a measure of the capacity of the muscle to gain or lose muscle mass.
Time Frame: 3 Months
Population: Maintenance hemodialysis (>3 months)
Measure: Mean (Standard Deviation); unit: Percentage of type 1 fibers
Groups:
- Exercise: Subjects will participate in a hybrid, center-based and home exercise training program for 3 months.
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 15
Percentage of type 1 fibers | 33.2 (11) | 30.0 (9)

3. Secondary Outcome: Quality of Life Score
Description: Disease-specific quality of life instrument is used to quantify broad quality of life domains, including physical function.
  Higher scores mean better values using a 0-100 scale.
Time Frame: 3 months
Population: Chronic kidney disease on maintenance hemodialysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 15
score on a scale | 48.7 (25.6) | 60.0 (22.3)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Subjects were monitored for any adverse events related to exercise testing, training, blood draws, and biopsy procedures. There were no adverse events during the study.
Arm/Group | Exercise | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT01990495/Prot_SAP_000.pdf